CLINICAL TRIAL: NCT05083858
Title: Comparison the Effectiveness of Cervical Stabilization and Oculomotor Exercises in Addition to the Classical Physiotherapy on Pain Severity, Joint Position Sense and Physical Parameters in Individuals With Chronic Neck Pain
Brief Title: Effect of Cervical Stabilization and Oculomotor Exercises on Position Sense With Chronic Neck Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Eastern Mediterranean University (Other)
Collaborators: Hacettepe University (Other)
Responsible Party: Principal Investigator, Cemaliye Hürer, Master of Science, Physiotherapist, Lecturer, Principal Investigator, Eastern Mediterranean University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HU
Record Dates: First submitted 2021-09-27; First posted 2021-10-19 (Actual); Last update posted 2021-10-19 (Actual); Status verified 2021-10

CONDITIONS: Chronic Neck Pain; Exercise Addiction
Keywords: Chronic Neck Pain; Proprioseption; Exercise; Stabilization; Oculomotor
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Classical Physiotherapy Program + Cervical Stabilization Exercises (Experimental): In addition to classical physiotherapy, Cervical Stabilization Exercises will be applied to the individuals in the 1st group.
  Interventions: Other: Classical Physiotherapy Program + Cervical Stabilization Exercises
- Classical Physiotherapy Program + Oculomotor Exercises (Experimental): In addition to classical physiotherapy, Oculomotor Exercises will be applied to the individuals in the 2nd group.
  Interventions: Other: Classical Physiotherapy Program + Oculomotor Exercises
- Classical Physiotherapy Program (Active Comparator): Only the classical physiotherapy program will be applied to the individuals in 3rd group.
  Interventions: Other: Classical Physiotherapy Program

INTERVENTIONS:
Other: Classical Physiotherapy Program + Cervical Stabilization Exercises — First of all, patients will be taught correct craniocervical flexion movement without activation of superficial muscles in different positions (supine, prone, crawling, sitting, standing). The program will be continued by asking to maintain the cranio-cervical flexion position during all movements. In order to gain dynamic stabilization, unilateral, bilateral, contralateral, ipsilateral and reciprocal extremity movements will be added to the program together with craniocervical flexion movement. Resistance will be added to the exercises as control of the movement is achieved. The exercises will progress from static to dynamic, from stationary floors to moving floors, from simple movements to complex movements.
  Other Names: Cervical Stabilization
  Arms: Classical Physiotherapy Program + Cervical Stabilization Exercises
Other: Classical Physiotherapy Program + Oculomotor Exercises — Oculomotor Exercises is a program consisting of exercises that support proprioception in the cervical region. It consists of 4 main contents; Sacadic Eye movements, Gaze stability, Head/eye coordination, Head repositioning exercise.
  Other Names: Oculomotor Exercises
  Arms: Classical Physiotherapy Program + Oculomotor Exercises
Other: Classical Physiotherapy Program — Conventional TENS will be applied to apply analgesic current. TENS application will be made to the cervical paravertebral region, using four 5 x 5 cm adhesive surface electrodes, at 80 Hz frequency for 20 minutes, 100 msec.
  All participants will be asked to lie in a prone position. The neck will be in a neutral position. The hot pack will be applied to the cervical region for 20 minutes.
  Classical massage will be applied for 20 minutes using the Swedish technique. The technique will be performed on the upper and neck region of the back with 3 strokes, 3 kneading and 3 strokes. The patient will be massaged while lying in the prone position.
  Stretching/Posture Exercises Exercises will be applied as a 5-10 minute warm-up-cool-down program at the beginning and end of the study. Cervical flexor, lateral flexor, rotator muscles, pectorals, inferior shoulder joint capsule will be stretched. In addition to this, posture exercises will also be done.
  Other Names: Classical Physiotherapy
  Arms: Classical Physiotherapy Program

SUMMARY:
The aim of this study is to compare the effectiveness of Cervical Stabilization and Oculomotor Exercises in addition to the classical physiotherapy on pain severity, cervical joint position sense, posture, cervical joint range of motion, strength and endurance of deep cervical flexor muscles, static and dynamic balance, neck awareness, functional disability and patient satisfaction in individuals with chronic neck pain. When the literature is examined, there is no study comparing the effectiveness of cervical stabilization and oculomotor exercises in individuals with chronic neck pain. However, it has also attracted our attention that a progressive and dynamic program was not followed in studies stating the oculomotor exercise program. In this sense, The study is important in terms of both comparing the effects of these 3 treatments and presenting a progressive and dynamic exercise protocol to the literature.

DETAILED DESCRIPTION:
The Participants included in the study will be divided into 3 groups. Participants in Group 1 will receive cervical stabilization exercises in addition to the classical physiotherapy program, individuals in Group 2 will receive oculomotor exercises in addition to the classical physiotherapy program, and only the classical physiotherapy program will be applied to group 3.

Transcutaneous Electrical Nerve Stimulation, hotpack, classical massage and stretching/posture exercises will be given to participants within the scope of the Classical Physiotherapy program. In addition to the classical physiotherapy program, the participants in the 1st and 2nd groups will be given exercises that gradually increase in difficulty level, 3 days a week, for a total of 8 weeks, under the control of a physiotherapist. Participants in the 3rd group will be given only classical physiotherapy. At the same time, stretching and posture exercises will be performed under the control of a physiotherapist.

ELIGIBILITY:
Inclusion Criteria:

* Men and women between the ages of 30-55,
* Neck pain for at least 3 months,
* Sedentary or non-regular exercise habit (3 days a week, less than 30 min of physical activity per day)
* According to the Numerical Pain Scale, the pain intensity is 4 cm and above

Exclusion Criteria:

* • Has received any physiotherapy program due to neck or back pain in the last 6 months,

  * Congenital anomaly in the cervical region (such as Klippel Feil Syndrome)
  * Having structural scoliosis at any level of the vertebral column,
  * Acute or chronic neurological deficits (sensory and motor loss),
  * With vertebrobasillary artery failure,
  * Thoracic Outlet Syndrome,
  * Any vestibular problem,
  * With marked diplopia and oculomotor muscle insufficiency,
  * Having a cervical rib,
  * Having a history of fractures in the cervical vertebrae,
  * Colorblind,
  * Suffering from whiplash injury,
  * Those with serious rheumatic diseases such as Ankylosing Spondylitis, Rheumatoid Arthritis
  * Having undergone spine surgery from any region,
  * Tumor or spinal cord compression due to another reason,
  * Using any pain reliever drug other than simple analgesics.
  * Those who have problems related to the lumbar region such as lumbal stenosis, lumbar disc herniation

Ages: 30 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 72 (Estimated)
Dates: Start 2021-08-01 (Actual); Primary Completion 2021-09-25 (Actual); Study Completion 2022-07 (Estimated)

PRIMARY OUTCOMES:
Cervical Joint Position Sense | Change from Cervical Joint Position Sense at the end of 8 weeks
  Joint Position Sense of flexion-extension, right-left rotation and right-left lateral flexion movements of the cervical region will be evaluated. A laser marker will be used to perform the assessment. The target angle for cervical flexion, extension and right-left rotation joint position sense measurement is 30°, and 20° for right-left cervical lateral flexion. Measurements will be made with eyes open and eyes closed. Before the JPS evaluations, the method will be explained to the individuals in detail and a sufficient number of trials will be made before the tests. Considering that fatigue may affect the results, all individuals will be warned not to forcefully move their neck and back muscles before the measurement. In order to prevent proprioceptive input, they will be asked to come in comfortable clothes that do not wrap around the neck on the day of their evaluation.

SECONDARY OUTCOMES:
Pain Intensity | Change from Pain Intensity at the end of 8 weeks
  Numerical Pain Scale will be used to determine the severity of neck pain at rest and during activity.An increase in the score means an increase in the severity of the patient's neck pain.
Craniovertebral Angle | Change from Craniovertebral Angle at the end of 8 weeks
  The posture of the cervical region will be evaluated by the lateral photographing method. Markers will be placed on specific anatomical points (C7, Tragus) and the lateral projections of these points will be used for angular calculations. The photos transferred to the computer will be transferred to the paint program and the lines connecting the markers will be drawn. Craniovertebral angle will be calculated using a computer program (Markus Bader-MB Software Solutions, Triangular Screen Ruler). Degree(°) is going to be record.
Cervical Joint Range of Motion | Change from Cervical Joint Range of Motion at the end of 8 weeks
  Inclinometer (Baseline Bubble Inclinometer) will be used to evaluate the joint range of motion of the cervical region. Measurements of cervical flexion, extension and right-left lateral flexion will be made in sitting position, and right and left rotation measurements will be made in supine position.
Strength and Endurance of the Deep Cervical Flexor Muscles | Change from Strength and Endurance of the Deep Cervical Flexor Muscles at the end of 8 weeks
  Craniocervical flexion test (CCFT) is used to evaluate the activation and static endurance of the deep flexor muscles of the cervical region. The test will be performed using Stabilizer Pressure Biofeedback (Chattanooga Stabilizer). The patient will be positioned in the supine position, with the cervical region in neutral position and the biofeedback pressure unit will be placed in the suboccipital space. The pressure cell will be inflated to 20 mmHg. Then, the individual will be instructed to perform a posterior tilt movement by increasing the pressure at 5 different levels (22, 24, 26, 28 and 30 mmHg.), Following the monitor of the device. After teaching the movement, the person will be asked to perform 10 contractions lasting 10 seconds at each level. The person will move to the next level after each successful attempt.
Static Balance | Change from Static Balance at the end of 8 weeks
  Stork balance test will be used in the evaluation of static balance. While one side is standing on one foot, the individual places the other foot on the inside of the knee on which she/he is standing. She/he places his hands on the waist and, with the signal of the physiotherapist, raises the heel of the supporting leg from the ground. She/he tries to maintain this position as long as he can stand with his eyes open . After the trial, She/he will be told to take this position three times with his eyes open and the holding times will be recorded. The best score of the recorded times will be taken.
Dynamic Balance | Change from Dynamic Balance at the end of 8 weeks
  It will be evaluated using the Y balance test. The reach distance in the anterior, posteromedial and posterolateral transport directions will be recorded. People will be asked to reach the furthest point with the other foot while trying to maintain balance with the dominant foot on the wooden platform while the hands are on the waist. 3 repetitions of reaching out in 3 directions will be recorded.
Neck Awareness | Change from Neck Awareness at the end of 8 weeks
  The Fremantle Neck Awareness Questionnaire will be used to assess neck awareness. Fremantle Neck Awareness Questionnaire is a 9-item questionnaire that evaluates neck perception, attention and proprioceptive awareness of individuals with chronic neck pain. The first 3 questions of the questionnaire, which evaluates awareness in 4 dimensions, evaluate attention, the fourth and fifth questions evaluate proprioceptive perception, and the sixth, seventh and ninth questions evaluate how the neck is perceived as shape and size relative to its body. The eighth question was interpreted as 'negligence'. The questions of the Likert-type questionnaire are between 0 and 4 points, meaning 0=Never, 1=Rarely, 2=Sometimes, 3=Often, 4=Always. The total score is 36. A high score indicates decreased awareness of the neck.
Functional Disability | Change from Functional Disability at the end of 8 weeks
  The Neck Disability Index (BDI) will be used to evaluate the functional disability of the neck. The questionnaire assesses how much neck pain associated with problems in the cervical region affects the individual in daily life and how much it interferes with the individual's daily work. The index consists of 10 items, 4 items evaluating subjective symptoms such as pain intensity, headache, concentration, sleep, and 6 items evaluating daily life activities such as personal care, lifting loads, reading, working life, driving, and leisure activities. Scoring is done between 0-5. The individual is asked to mark the answer that best fits him. If the total score obtained in the index is between 0-4, it is classified as no disability, between 5-14 as mild disability, between 15-24 as moderate disability, between 25-34 as severe disability and above 35 points as total disability.
Patient Satisfaction | End of eight weeks
  The Global Perceived Impact (GAE) questionnaire will be used to assess the extent to which individuals benefit from treatment after treatment. This questionnaire is used to evaluate the extent to which individuals benefit from treatment after treatment. Individuals are asked to rate between 1 (very much improved) and 9 (very much worsened) to the question 'How have your complaints changed compared to the time before your treatment?'. Scale scores were, in order, 1-very much improved, 2-very much improved, 3-moderately improved, 4-slightly improved, 5-unchanged, 6-slightly worsened, 7-moderately worsened, 8-very much worsened, 9-very much worsened. is in the form. Scoring will be done once at the end of the treatment.
Cervicothoracic angle | Change from Cervicothoracic angle at the end of 8 weeks
  The posture of the cervical region will be evaluated by the lateral photographing method. Markers will be placed on specific anatomical points (C7, Tragus and T4) and the lateral projections of these points will be used for angular calculations. The photos transferred to the computer will be transferred to the paint program and the lines connecting the markers will be drawn. Cervicothoracic angle will be calculated using a computer program (Markus Bader-MB Software Solutions, Triangular Screen Ruler). Degree(°) is going to be record.

CONTACTS AND LOCATIONS:
Overall Officials: Zafer Erden, Principal Investigator — Hacettepe University
Locations (1):
- Eastern Mediterranean University, Famagusta, Cyprus

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jull GA, Falla D, Vicenzino B, Hodges PW. The effect of therapeutic exercise on activation of the deep cervical flexor muscles in people with chronic neck pain. Man Ther. 2009 Dec;14(6):696-701. doi: 10.1016/j.math.2009.05.004. Epub 2009 Jul 25. PMID 19632880
- [Background] Revel M, Minguet M, Gregoy P, Vaillant J, Manuel JL. Changes in cervicocephalic kinesthesia after a proprioceptive rehabilitation program in patients with neck pain: a randomized controlled study. Arch Phys Med Rehabil. 1994 Aug;75(8):895-9. doi: 10.1016/0003-9993(94)90115-5. PMID 8053797
- [Background] Jull G, Falla D, Treleaven J, Hodges P, Vicenzino B. Retraining cervical joint position sense: the effect of two exercise regimes. J Orthop Res. 2007 Mar;25(3):404-12. doi: 10.1002/jor.20220. PMID 17143898
- [Background] Strimpakos N, Sakellari V, Gioftsos G, Kapreli E, Oldham J. Cervical joint position sense: an intra- and inter-examiner reliability study. Gait Posture. 2006 Jan;23(1):22-31. doi: 10.1016/j.gaitpost.2004.11.019. PMID 16311191